CLINICAL TRIAL: NCT02813785
Title: A Phase III, Open-Label, Multicenter, Randomized Study to Investigate the Efficacy and Safety of Atezolizumab (Anti-PD-L1 Antibody) Compared With Docetaxel in Patients With Non-Small Cell Lung Cancer After Failure With Platinum-Containing Chemotherapy
Brief Title: A Study of Atezolizumab Compared With Docetaxel in Non-Small Cell Lung Cancer (NSCLC) After Failure With Platinum-Containing Chemotherapy
Acronym: IMpower210
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: YO29232
Record Dates: First submitted 2016-06-23; First posted 2016-06-27 (Estimated); Last update posted 2023-01-10 (Actual); Status verified 2023-01

CONDITIONS: Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — atezolizumab; Docetaxel

ARMS (2):
- Atezolizumab (Experimental): Participants will receive atezolizumab until loss of clinical benefit and will thereafter enter survival follow-up until death, loss to follow-up, withdrawal, or study end.
  Interventions: Drug: Atezolizumab (MPDL3280A), an engineered anti-PD-L1 antibody
- Docetaxel (Active Comparator): Participants will receive docetaxel until disease progression per standard RECIST v1.1 criteria or unacceptable toxicity and will thereafter enter survival follow-up until death, loss to follow-up, withdrawal, or study end.
  Interventions: Drug: Docetaxel

INTERVENTIONS:
Drug: Atezolizumab (MPDL3280A), an engineered anti-PD-L1 antibody — Atezolizumab will be administered at a fixed dose of 1200 milligrams (mg) via intravenous (IV) infusion on Day 1 of each 21-day cycle.
  Other Names: MDPL3280A, RO5541267
  Arms: Atezolizumab
Drug: Docetaxel — Docetaxel will be administered as 75 milligrams per square meter (mg/m^2) via IV infusion on Day 1 of each 21-day cycle.
  Other Names: Taxotere
  Arms: Docetaxel

SUMMARY:
This Phase III, multicenter, open-label, randomized, controlled study is designed to evaluate the efficacy and safety of the anti-programmed death-ligand 1 (PD-L1) antibody atezolizumab compared with docetaxel in participants with locally advanced or metastatic NSCLC who have progressed during or following a platinum-containing regimen. Treatment may continue until disease progression, loss of clinical benefit, or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Histologically documented, locally advanced or metastatic NSCLC
* Representative formalin-fixed paraffin-embedded (FFPE) tumor specimens available or at least 12 unstained, freshly cut serial sections with associated pathology report that are evaluable for PD-L1 expression and epidermal growth factor receptor (EGFR) mutation status prior to enrollment, except for known sensitizing EGFR mutations in which case 10 unstained slides are required and there is no need for central testing of EGFR mutation status
* Disease progression during or following treatment with a prior platinum-containing regimen for locally advanced, unresectable, inoperable, or metastatic NSCLC, or disease recurrence within 6 months of treatment with a platinum-based adjuvant and/or neoadjuvant regimen or combined modality with curative intent
* Measurable disease per RECIST v1.1
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Life expectancy greater than or equal to (>/=) 12 weeks
* Adequate hematologic and end organ function
* Agreement to remain abstinent or use contraceptive methods among women of childbearing potential or male partners of women of childbearing potential
* Recovery from all acute toxicities from previous therapy

Exclusion Criteria:

* Active or untreated central nervous system (CNS) metastases
* Spinal cord compression not definitively treated or not clinically stable
* Leptomeningeal disease
* Uncontrolled pleural or pericardial effusions or ascites requiring recurrent drainage
* Uncontrolled tumor-related pain
* Uncontrolled hypercalcemia
* Malignancies other than NSCLC within 5 years prior to randomization, except for those curatively treated with negligible risk of metastasis or death
* Pregnant or lactating women
* Significant cardiovascular, pulmonary, or autoimmune disease
* Severe infection or major surgery within 4 weeks, or antibiotic treatment within 2 weeks prior to randomization
* Prior treatment with or hypersensitivity to study drug(s) or related compounds
* Inability to discontinue strong cytochrome P450 (CYP) 3A4 inhibitors
* Prior allogeneic bone marrow or solid organ transplant
* Known PD-L1-negative expression status
* Positive human immunodeficiency virus (HIV) or active hepatitis B or C
* Receipt of a live attenuated vaccine within 4 weeks prior to randomization
* Treatment with systemic immunomodulators within 4 weeks or five half-lives (whichever is shorter) prior to randomization
* Treatment with systemic corticosteroids within 2 weeks prior to randomization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 565 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2022-12-27 (Actual)

PRIMARY OUTCOMES:
Overall Survival (OS) | Baseline until death from any cause (up to approximately 3 years)

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) According to Response Evaluation Criteria in Solid Tumors (RECIST) Version (v) 1.1 | Baseline until disease progression or death from any cause (up to approximately 3 years)
Percentage of Participants with Objective Response According to RECIST v1.1 | Baseline until disease progression or death from any cause (up to approximately 3 years)
Duration of Objective Response According to RECIST v1.1 | From first objective response until disease progression or death from any cause (up to approximately 3 years)
Percentage of Participants with Adverse Events | From start of treatment until 90 days after treatment discontinuation or initiation of other anti-cancer therapy (up to approximately 3 years)
Percentage of Participants with Anti-Therapeutic Antibodies (ATAs) to Atezolizumab | Predose (0 hours) on Day 1 of Cycles 1, 2, 3, 4, 8, 16, and every eight cycles thereafter (cycle length of 21 days) until/at treatment discontinuation (up to approximately 3 years) and 120 days after last dose (up to approximately 3 years overall)
Minimum Observed Serum Concentration (Cmin) of Atezolizumab | Predose (0 hours) on Day 1 of Cycles 1, 2, 3, 4, 8, 16, and every eight cycles thereafter (cycle length of 21 days) until/at treatment discontinuation (up to approximately 3 years) and 120 days after last dose (up to approximately 3 years overall)
Time to Deterioration (TTD) in Lung Cancer Symptoms According to European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ) Core 30 C30) | From start of treatment until treatment discontinuation (up to approximately 3 years)
TTD in Lung Cancer Symptoms According to EORTC QLQ Lung Cancer Module (LC13) | From start of treatment until treatment discontinuation (up to approximately 3 years)
Health-Related Quality of Life According to EORTC QLQ-C30 Score | Day 1 of every cycle (cycle length of 21 days) until/at treatment discontinuation (up to approximately 3 years)
Health-Related Quality of Life According to EORTC QLQ-LC13 Score | Day 1 of every cycle (cycle length of 21 days) until/at treatment discontinuation (up to approximately 3 years)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (38):
- China (26):
  - Cancer Hospital Chinese Academy of Medical Sciences., Beijing
  - Beijing Cancer Hospital, Beijing
  - Beijing Chest Hospital; Oncology Department, Beijing
  - Affiliated Hospital of Bengbu Medical College, Bengbu
  - the First Hospital of Jilin University, Changchun
  - Jilin Cancer Hospital, Changchun
  - Changzhou First People's Hospital, Changzhou
  - West China Hospital, Sichuan University, Chengdu
  - Second Affiliated Hospital of Third Military Medical University, Chongqing
  - Third Affiliated Hospital of Third Military Medical University, Chongqing
  - Guangdong General Hospital, Guangzhou
  - The First Affiliated Hospital of Guangzhou Medical University, Guangzhou
  - Sun Yet-sen University Cancer Center, Guangzhou
  - The First Affiliated Hospital of College of Medicine, Zhejiang University, Hangzhou
  - Sir Run Run Shaw Hospital, Hangzhou
  - Harbin Medical University Cancer Hospital, Harbin
  - Jiangsu Cancer Hospital, Nanjing
  - The Affiliated Hospital of Medical College Qingdao University, Qingdao
  - Shanghai chest hospital, Shanghai
  - Zhongshan Hospital Fudan University, Shanghai
  - Fudan University Shanghai Cancer Center, Shanghai
  - Liaoning cancer Hospital & Institute, Shenyang
  - Tianjin Medical University General Hospital, Tianjin
  - The First Affiliated Hospital of Xian Jiao Tong University, Xi'an
  - Zhejiang Cancer Hospital, Zhejiang
  - Henan Cancer Hospital, Zhengzhou
- Malaysia (3):
  - Sarawak General Hospital; Department of Radiotherapy, Oncology and Palliative care, Sarawak, Sarawak
  - Hospital Sultan Ismail; Oncology, Johor Bahru
  - Hospital Kuala Lumpur; Jabatan Radioterapi dan Onkologi, Kuala Lumpur
- National Cancer Centre; Medical Oncology, Singapore, Singapore
- South Korea (4):
  - Kyungpook National University Medical Center, Daegu
  - Chungnam National University Hospital, Daejeon
  - Chonnam National University Hwasun Hospital, Jeollanam-do
  - Korea University Guro Hospital, Seoul
- Thailand (4):
  - Chulalongkorn Hospital; Medical Oncology, Bangkok
  - Ramathibodi Hospital; Dept of Med.-Div. of Med. Onc, Bangkok
  - Faculty of Med. Siriraj Hosp.; Med.-Div. of Med. Oncology, Bangkok
  - CHIANG MAI UNI HOSPITAL; FACULTY OF MEDICINE; Medical Oncology unit, Chiang Mai